CLINICAL TRIAL: NCT05171179
Title: A Prospective, Randomized Controlled Trial Investigating Pecs Blocks Types I and II as a Method for Administering the Non-Opioid Anesthetic Exparel in Order to Mitigate Postoperative Narcotic Usage, Pain, Nausea, and Hospital Stay in Patients Undergoing Implant-Based Tissue Expander Breast Reconstruction Surgery
Brief Title: The Use of Pecs Blocks in Combination With Exparel in Breast Reconstruction Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Robert Galiano, Associate Professor of Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00214187
Record Dates: First submitted 2021-11-04; First posted 2021-12-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-02

CONDITIONS: Mammaplasty
Keywords: breast reconstruction; mammaplasty; analgesic
MeSH Terms: interventions — Mammaplasty; Bupivacaine

STUDY DESIGN:
Intervention Model Description: 1. Group 1: Use of Pecs block types I and II with bupivacaine as local anesthetic
  2. Group 2: Use of Pecs block types I and II with mixture of bupivacaine and Exparel* (*Must include bupivacaine at lower dose to decrease intra-operative variability in pain control due to delayed onset of Exparel and in ability to use lidocaine infusion with injection of Exparel)
Who Masked: Participant
Masking Description: Patient will be randomized into one of the two trial arms. Randomization process will involve 60 envelopes, 30 of which will contain assignment to the study arm with Exparel blocks and 30 which will contain assignment to bupivacaine blocks. The PI's attending nurse will randomly distribute an envelope to the study team between V1 and V2. V2, the day of surgery, will be the only visit where the patient would potentially have contact with the treatments. The patient will not be aware of what treatment they receive until after their 2-week follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blocks+Bupivacaine (Active Comparator): Use of Pecs block types I and II with bupivacaine as local anesthetic
  Interventions: Procedure: Breast Reconstruction (Mammaplasty); Device: Pecs blocks; Drug: Bupivacaine
- Blocks+Bupivacaine+Exparel (Experimental): Use of Pecs block types I and II with mixture of bupivacaine and Exparel* (*Must include bupivacaine at lower dose to decrease intra-operative variability in pain control due to delayed onset of Exparel)
  Interventions: Procedure: Breast Reconstruction (Mammaplasty); Device: Pecs blocks; Drug: Exparel; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Breast Reconstruction (Mammaplasty) — Breast Reconstruction (mammaplasty) surgery with implant-based tissue expander
Device: Pecs blocks — Pectoral nerve (Pecs) blocks I and II function by blocking the pectoral, intercostal, intercostobrachial nerves, and/or long thoracic nerve. These are used primarily for breast surgeries and are gaining momentum as simple administers of local analgesics. Pecs blocks utilize ultrasound to guide injection of local analgesic. It is less invasive and more accurate than most current modes of analgesia administration.
  Other Names: Pecs blocks I and II
Drug: Exparel — Exparel is a sterile, non-pyrogenic white to off-white preservative-free aqueous suspension of multivesicular liposomes (DepoFoam® drug delivery system) containing bupivacaine. Bupivacaine is present at a concentration of 13.3 mg/mL. After injection of Exparel, bupivacaine is released from the multivesicular liposomes over a period of time.
  Arms: Blocks+Bupivacaine+Exparel
Drug: Bupivacaine — This is an anesthetic delivered during breast reconstruction surgery that will be given to participants in both arms.

SUMMARY:
This project intends to more thoroughly investigate the direct influence of Pecs blocks in the administration of Exparel, a non-opioid analgesic, in breast reconstruction surgery. The hypothesis is that this analgesic delivery method will significantly reduce negative outcomes such as post-operative pain, opioid use, and nausea while increasing positive outcomes such as post-operative physical activity.

DETAILED DESCRIPTION:
The research team will be investigating the use of a novel type of local drug administration as well as assessing whether a non-opioid based drug will result in more positive pain outcomes while reducing reliance on narcotics (opioid-based drugs) following surgery.

The drug administration tool, called the Pecs blocks types I and II, utilizes ultrasound to help guide anesthetic injection for local anesthesia. This has been an effective way to deliver local anesthetic during breast surgeries. Meanwhile, a non-opioid analgesic drug (similar to an anesthetic, meaning it is used during surgery to reduce pain) called Exparel has been shown to reduce post-operative use of narcotics, length of stay in hospitals, and pain compared to the current standards in breast reconstruction surgery. Exparel is approved by the FDA for use in surgical sites during breast reconstruction surgery. Exparel has shown to reduce pain and post-surgical nausea and vomiting in breast reconstruction patients. However, the combination of Exparel with Pecs blocks has not been examined in breast reconstruction surgery, and the research team suspects that breast reconstruction patients who are administered Exparel with Pecs blocks will experience less pain, increased mobility, and less nausea following surgery. Furthermore, the researchers believe that this non-opioid based drug could reduce the necessity to use narcotics following surgery. Narcotics are highly addictive and can lead to dependency following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects greater than 18 years of age.
2. Subject who are undergoing implant-based, tissue expander breast reconstruction surgery.

Exclusion Criteria:

1. Subjects undergoing flap breast reconstruction.
2. Subjects who are undergoing direct-to-implant surgery.
3. Subjects who have previously undergone radiation therapy.
4. Medical or psychiatric condition that may increase the risk associated with study participation, may complicate patient compliance, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
5. Subjects who are pregnant at the date of surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 2 weeks post op
  • Investigate amount of post-operative opioid consumption post operatively

SECONDARY OUTCOMES:
Nausea | 2 weeks post op
  • Assess Post-Operative Nausea scores between the two arms using the participant-recorded Edmonton Symptom Assessment tool which scores on a scale of one to ten, where ten is the most nausea experienced
Mobility | 2 weeks post op
  • Assess post-operative mobility using the participant-recorded Edmonton Symptom Assessment tool which scores on a scale of one to ten where ten is the most immobile
Pain Outcomes | 2 weeks post op
  • Assess the pain patients experience throughout their recovery period using the participant-recorded Edmonton Symptom Assessment tool which scores on a scale of one to ten where ten is the highest pain

CONTACTS AND LOCATIONS:
Overall Officials: Robert Galiano, MD, Principal Investigator — 3126956022
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No